CLINICAL TRIAL: NCT03938805
Title: Internet-based Cognitive Behavioural Therapy Program Tailored to Patients With Cardiovascular Disease and Insomnia - Effects of a Randomised Controlled Trial
Brief Title: I-CBT Tailored to Patients With Cardiovascular Disease and Insomnia
Acronym: Hit-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonkoping University (Other)
Responsible Party: Principal Investigator, Anders Broström, Professor, Jonkoping University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/258-31
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Insomnia; Cardiovascular Diseases
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. The intervention group participated in a nine-week internet-based cognitive behavioral therapy program. The initial parts of the program, focusing on cardiovascular disease was initially tailored to fit patients with heart failure and has undergone pilot testing. The intervention program used in the current study was adapted to fit also patient with other cardiovascular diagnoses (i.e., heart failure, myocardial infarction, atrial fibrillation) and comprise 1-week of introduction, 2 weeks psycho education on cardiovascular diseases/insomnia, 6 weeks of sleep hygiene, stimulus control and sleep restriction. The Control Group receive 3 weeks of internet-based sleep hygiene education.
Who Masked: Investigator
Masking Description: Single blinded (PI). The randomization is performed by a study team member who was blinded to screening and baseline data. The physician who assessed the patients had access to them in a random sequence. Patients were randomized 1.1 to nine-week internet-based cognitive behavioral therapy (intervention group) or online 3 weeks sleep hygiene (control group) generated by an independent researcher using a block size of two. Masking of patients was not possible since the interventions is a internet-based cognitive behavioral therapy program. Outcome measures were not necessary to mask since these were automatically collected via the study platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CBT (Experimental): Internet-based cognitive behavioral therapy program including 1-week introduction, 2 weeks psycho education on Cardiovascular disease/insomnia, 6 weeks of sleep hygiene, stimulus control and sleep restriction
  Interventions: Behavioral: Internet-based cognitive behavioral therapy for insomnia
- Control group (Active Comparator): 3 weeks internet-based sleep hygiene education
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy for insomnia — Patients will be provided with psycho education on different cardiovascular diseases, sleep, insomnia, and provided with different behavioral techniques to improve their sleep. The participants in the intervention Group who receives the Internet-based cognitive behavioral therapy program will also have access to support given by a nurse specialized in sleep. A module is given each week during the 9-week intervention.
  Other Names: Internet-based CBT
  Arms: I-CBT
Other: Control group — Control group receiving 3 weeks internet-based education on sleep hygiene. A module is given each week during the 3 weeks.
  Arms: Control group

SUMMARY:
The Hit-IT study is based on an internet-based cognitive behavioral therapy program tailored to patients with different types of cardiovascular diseases and insomnia. A randomized controlled trial design is used. A 9 weeks internet-based cognitive behavioral therapy intervention vs a 3 weeks sleep hygiene education.

DETAILED DESCRIPTION:
DESIGN: Randomized controlled trial with 1-year follow-up. All patients with cardiovascular disease (i.e., myocardial infarction, heart failure, atrial fibrillation and angina) from 4 primary care centers will be screened for insomnia and during a clinical examination diagnosed by a physician specialized in sleep medicine. INTERVENTION: 9 weeks internet-based cognitive behavioral therapy for insomnia (1 week introduction, 2 weeks psycho education on cardiovascular disease/insomnia, 6 weeks of sleep hygiene, stimulus control and sleep restriction) vs 3 weeks internet-based sleep hygiene education. QUESTIONNAIRES: Sleep (Pittsburgh Sleep Quality Index, Insomnia Severity Index, sleep diary), depressive- and cardiac symptoms (Patient Health Questionnaire-9, Cardiac Anxiety Questionnaire) and Quality of Life (SF-12) at baseline, during and after intervention (after 6 and 12 months).

ELIGIBILITY:
Inclusion criteria:

* age over 18 years
* having a clinical diagnose of insomnia
* being treated for heart failure, coronary artery disease or atrial fibrillation
* access to a computer with an Internet connection, access to a mobile phone and was willing to participate in a treatment for their insomnia.

Exclusion criteria:

* no access to internet, computer or cellphone.
* not understanding the Swedish language
* suffering from cognitive disabilities, severe psychiatric disease, severe somatic disease or sleep apnea
* suffering from drug abuse
* been hospitalised for heart failure, coronary artery disease or atrial fibrillation in the last four weeks
* expected survival less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Insomnia severity index (ISI) | 12 months
  The Insomnia severity index is a self-assessment questionnaire that measure the perceived severity of insomnia symptoms such as, falling asleep, staying asleep, numbers of awakenings, early awakening, sleep satisfaction. The scale includes of seven items, scored on a 0- 4 scale that are summed to a range of 0 - 28. The score can be divided into four categories: no clinical insomnia (0-7), subthreshold insomnia (8-14), clinical insomnia of moderate severity (15-21), and severe clinical insomnia (22-28). The total score and the categories will be used.

SECONDARY OUTCOMES:
Short Form 12 (SF-12) | 12 months
  The Short Form 12 Health Survey is a self-assessment questionnaire that measures the respondents quality of life through 12 questions. The 12 items are rated on a 5-point Likert scale, and 2 component scale scores (i.e., the physical component scale and the mental component scale) will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Broström, Professor, Principal Investigator — Jonkoping University
Locations (1):
- Jönköping University, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Sleep (Pittsburg Sleep Quality Index, Insomnia Severity Index, sleep diary), depressive- and cardiac symptoms (Patient Health Qurestionnaire-9, Cardiac Anxiety Questionnaire) and Quality of Life (SF-12) at baseline, during and after intervention (after 6 and 12 months).

REFERENCES:
- [Derived] Siebmanns S, Johansson P, Ulander M, Johansson L, Andersson G, Brostrom A. The effect of nurse-led Internet-based cognitive behavioural therapy for insomnia on patients with cardiovascular disease: A randomized controlled trial with 6-month follow-up. Nurs Open. 2021 Jul;8(4):1755-1768. doi: 10.1002/nop2.817. Epub 2021 Feb 20. PMID 33609425